CLINICAL TRIAL: NCT01317914
Title: Epidemiology of Celiac Disease: A Prospective Study of Undiagnosed Celiac Disease in the Community
Brief Title: Prospective Study of Undiagnosed Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph A. Murray, M.D., Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-000178
Record Dates: First submitted 2010-09-23; First posted 2011-03-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary instruction on Gluten Free Diet (Experimental)
  Interventions: Other: Dietary instruction

INTERVENTIONS:
Other: Dietary instruction — Subjects subsequently diagnosed with celiac disease will have gluten-free diet instructions given by registered dietitian experienced in the gluten-free diet. Subjects will have follow-up in 3 months time from initial instruction to verify compliance.

SUMMARY:
Direct benefits to the participants, who are diagnosed with celiac disease may be substantial and could include lessening or prevention of GI symptoms, correction of biochemical abnormalities and reduction in risk for malignancies or bone disease which are most common in untreated celiac disease. However, the precise benefit is unknown and the motivation for this proposed study. If these individuals have a positive celiac serology test at the present time there is a high likelihood that they may have celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years old
* Male and female

Retrospective testing for celiac disease was done on previously stored serum. Contacting specific individuals for inclusion into study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Understanding the impact of undiagnosed celiac disease and the potential benefits of diagnosis | one year
  To understanding the impact of undiagnosed celiac disease and the potential benefits, detection and treatment may have a substantial impact on the health of these subjects and the large numbers of Americans with undiagnosed celiac disease. The outcome measures we will be looking at are Quality of Life, GI Symptoms including diarrhea, constipation, abdominal pain, Tissue Transglutaminase level improvement after 12 weeks on a gluten free diet, bone density, understanding of a gluten free diet.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States